CLINICAL TRIAL: NCT00309777
Title: Study of Pitavastatin Vs. Simvastatin (Following Up-Titration) in Patients With Primary Hypercholesterolemia or Combined Dyslipidemia
Brief Title: Study to Compare the Efficacy and Safety of Pitavastatin and Simvastatin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kowa Research Europe (Industry)
Responsible Party: Neil Hounslow, MD, Kowa Research Europe, Ltd.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NK-104-302; EudraCT number 2005-001033-15
Record Dates: First submitted 2005-11-11; First posted 2006-04-03 (Estimated); Results first posted 2009-12-16 (Estimated); Last update posted 2010-01-12 (Estimated); Status verified 2010-01

CONDITIONS: Hypercholesterolemia; Dyslipidemia
Keywords: hypercholesterolemia; kowa; dyslipidemia; pitavastatin; NK-104; Primary Hypercholesterolemia or Combined Dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — pitavastatin; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Pitavastatin 2 mg (Experimental): Pitavastatin 2 mg once daily
  Interventions: Drug: Pitavastatin
- Simvastatin 20 mg (Active Comparator): Simvastatin 20 mg once daily
  Interventions: Drug: Simvastatin
- Pitavastatin 4 mg (Experimental): Pitavastatin 4 mg once daily
  Interventions: Drug: Pitavastatin
- Simvastatin 40 mg (Active Comparator): Simvastatn 40 mg once daily
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin once daily
  Arms: Pitavastatin 2 mg; Pitavastatin 4 mg
Drug: Simvastatin — Simvastatin once daily
  Arms: Simvastatin 20 mg; Simvastatin 40 mg

SUMMARY:
The purpose of this study is to compare the efficacy and safety of pitavastatin with that of simvastatin.

ELIGIBILITY:
Inclusion Criteria:

* Males and females (18-75 years)
* Must have been following a restrictive diet
* Diagnosis of primary hypercholesterolemia or combined dyslipidemia

Exclusion Criteria:

* Homozygous familial hypercholesterolemia or familial hypoalphalipoproteinemia;
* Conditions which may cause secondary dyslipidemia.
* Uncontrolled diabetes mellitus (by hemoglobin A1c [HbA1c] > 8%)
* Abnormal serum creatine kinase (CK) above the pre-specified level
* Abnormal pancreatic, liver or renal function
* Significant heart disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 857 (Actual)
Dates: Start 2005-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dragos Budinski, Med Dr., Study Director — Medical Director
Locations (42):
- Finland (5):
  - Geri-Med Oy, Helsinki
  - Kaisaniemen Laakariasema, Helsinki
  - Keravan Laakarikeskus, Helsinki
  - SOK-tyoterveyshuolto, Tampere
  - TYKS University Hospital, Turku
- Italy (10):
  - Dipartimento Di Medicina Clinica e Biotecnologia Applicata, Bologna
  - Centro di Ricerca Clinica, Chieti
  - Gerontologia e Geriatria - Universita degli Studi, Ferrara
  - Dipartimento di Medicina Interna DIMI, Genova
  - Universita di Modena e Reggio Emilia, Policlinico, Modena
  - Dipartimento di Medicina Clinica e Sperimentale, Napoli
  - Medicina Clinica e delle Patologie Emergenti, Palermo
  - Dipartimento di Medicina Interna e Scienze Biomediche, Parma
  - U.O Malattie Metaboliche e Diabetologia, Treviglio
  - Azienda Ospedaliero-Universitaria, Trieste
- Norway (5):
  - Volvat Medisinske Senter, Fredrikstad
  - Nyomen Legekontor, Kongsberg
  - Radhuset Spesialistsenter, Oslo
  - Rikshospitalet - University Hospital, Oslo
  - Skedsmo Medisinske Senter A.S., Skedsmokorset
- Russia (12):
  - Kemerovo Cardiology Dispensary, Kemerovo
  - Central Clinical Hospital 1 of RZD, Moscow
  - City Clinical Hospital 23, Moscow
  - City Clinical Hospital 64, Moscow
  - Moscow City Clinical Hospital 68, Moscow
  - State Research Center for Preventive Medicine, Moscow
  - Novosibirsk Reg. Clinical Cardiology Dispensary, Novosibirsk
  - Central Medical Unit 122, St. Pb, Saint Petersburg
  - Clinical Hospital of Russian Academy of Sciences, Saint Petersburg
  - Consulting and Diagnostic Center 85, Saint Petersburg
  - Krestovsky Island Medical Institute, Saint Petersburg
  - Pokrovskaya City Hospital, Saint Petersburg
- United Kingdom (10):
  - St Michael's Partnership, Bath
  - Avondale Surgery, Chesterfield
  - Knowle House Surgery, Plymouth
  - The Burngreave Surgery, Sheffield
  - St Helier Hospital, Surrey
  - Box Surgery, Wiltshire
  - Eastleigh Surgery, Wiltshire
  - Lovemead Group Practice, Wiltshire
  - St Chad's Surgery, Wiltshire
  - The Health Centre, Wiltshire

REFERENCES:
- [Derived] Ose L, Budinski D, Hounslow N, Arneson V. Comparison of pitavastatin with simvastatin in primary hypercholesterolaemia or combined dyslipidaemia. Curr Med Res Opin. 2009 Nov;25(11):2755-64. doi: 10.1185/03007990903290886. PMID 19785568

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were randomized to one of 4 treatment arms based on inclusion/exclusion criteria.
Pre-assignment Details: After a 6-8 week run in period when no lipid lowering therapy was allowed, subjects were randomized to one of 4 treatment arms.
Period: Overall Study
Arm/Group | Pitavastatin 2 mg | Simvastatin 20 mg | Pitavastatin 4 mg | Simvastatin 40 mg
Started | 315 | 108 | 323 | 111
Safety Population | 311 (All randomized patients who received at least one dose of study treatment.) | 107 (All randomized patients who received at least one dose of study treatment.) | 320 (All randomized patients who received at least one dose of study treatment.) | 110 (All randomized patients who received at least one dose of study treatment.)
Completed | 292 | 99 | 304 | 107
Not Completed | 23 | 9 | 19 | 4
Not completed — Adverse Event | 13 | 2 | 8 | 1
Not completed — Protocol Violation | 4 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 6 | 5 | 7 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pitavastatin 2 mg | Simvastatin 20 mg | Pitavastatin 4 mg | Simvastatin 40 mg | Total
Number analyzed (Participants) | 311 | 107 | 320 | 110 | 848
Age, Categorical [Count of Participants; unit: Participants] — Data presented are for the safety population, defined as all randomized patients who receive at least one dose of the study drug.
  Participants
    <=18 years | 0 | 0 | 0 | 0 | 0
    Between 18 and 65 years | 214 | 72 | 231 | 76 | 593
    >=65 years | 97 | 35 | 89 | 34 | 255
Age Continuous [Mean (Standard Deviation); unit: years] — Data presented are for the safety population, defined as all randomized patients who receive at least one dose of the study drug.
  years | 58.7 (8.83) | 58.6 (9.64) | 57.7 (8.97) | 58.4 (9.54) | 58.3 (9.08)
Sex: Female, Male [Count of Participants; unit: Participants] — Data presented are for the safety population, defined as all randomized patients who receive at least one dose of the study drug.
  Participants
    Female | 196 | 63 | 195 | 48 | 502
    Male | 115 | 44 | 125 | 62 | 346

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low Density Lipoprotein-cholesterol (LDL-C) at 12 Weeks
Description: Percent change from baseline in low density lipoprotein-cholesterol (LDL-C)after 12 Weeks
Time Frame: Baseline to 12 weeks
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Pitavastatin 2 mg | Simvastatin 20 mg | Pitavastatin 4 mg | Simvastatin 40 mg
Number analyzed (Participants) | 307 | 107 | 319 | 110
Percent change | -38.99 (14.573) | -34.97 (15.528) | -43.97 (14.494) | -42.84 (15.769)

2. Secondary Outcome: National Cholesterol Education Program (NCEP) LDL-C Target Attainment
Description: Number of subjects achieving National Cholesterol Education Program (NCEP) LDL-C Target (LDL less than or equal to 130 mg/dL)at Week 12
Time Frame: 12 week
Population: Full Analysis Set
Measure: Number; unit: Participants
Arm/Group | Pitavastatin 2 mg | Simvastatin 20 mg | Pitavastatin 4 mg | Simvastatin 40 mg
Number analyzed (Participants) | 307 | 107 | 319 | 110
Participants | 215 | 69 | 253 | 86

ADVERSE EVENTS:
Arm/Group | Pitavastatin 2 mg | Simvastatin 20 mg | Pitavastatin 4 mg | Simvastatin 40 mg
Serious Adverse Events (participants affected / at risk) | 3/311 | 2/107 | 4/320 | 2/110
Other Adverse Events (participants affected / at risk) | 56/311 | 28/107 | 44/320 | 10/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 2 mg (N=311) | Simvastatin 20 mg (N=107) | Pitavastatin 4 mg (N=320) | Simvastatin 40 mg (N=110)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Pleuropericarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0
Sudden cardiac death (General disorders) | 0 | 1 | 0 | 0
Anaphylactic reation (Immune system disorders) | 1 | 0 | 0 | 0
Campylobacter intestinal infection (Infections and infestations) | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 2
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pitavastatin 2 mg (N=311) | Simvastatin 20 mg (N=107) | Pitavastatin 4 mg (N=320) | Simvastatin 40 mg (N=110)
Influenza (Infections and infestations) | 4 | 6 | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 1 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 3 | 7 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 3 | 6 | 3
Diarrhea (Gastrointestinal disorders) | 8 | 2 | 6 | 1
Nausea (Gastrointestinal disorders) | 4 | 3 | 6 | 1
Headache (Nervous system disorders) | 10 | 4 | 11 | 2
Fatigue (General disorders) | 7 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days